CLINICAL TRIAL: NCT04738565
Title: An Innovative Probiotic Product With Antiallergic Properties. The Effectiveness of a Mixture of Lactobacillus ŁOCK Strains in Children With Atopic Dermatitis - Multicentre, Randomized, Double-blind Placebo Controlled Trial.
Brief Title: An Innovative Probiotic Product With Antiallergic Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Memorial Health Institute, Poland (Other)
Responsible Party: Principal Investigator, Bożena Cukrowska, professor of medicine, MD, PhD, Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N R12-0101-10/2011
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Atopic Dermatitis; Food Allergy; Effects of Probiotics
MeSH Terms: conditions — Dermatitis, Atopic; Food Hypersensitivity | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): The mixture of 3 probiotic strains in the following proportions: 50% Lactobacillus casei ŁOCK 0919, 25% Lactobacillus rhamnosus ŁOCK 0908, 25% Lactobacillus rhamnosus ŁOCK 0900 (Latopic® preparation, Biomed S.A., Cracow, Poland).
  Interventions: Dietary Supplement: Probiotic preparation
- Maltodextrin (Placebo Comparator): Maltodextrin - a substance in which probiotic strains have been suspended.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic preparation — The mixture of Lactobacillus rhamnosus ŁOCK 0900, Lactobacillus rhamnosus ŁOCK 0908 and Lactobacillus casei ŁOCK 0919 administered once a day at a dose of one billion for 3 months.
  Arms: Probiotic
Dietary Supplement: Maltodextrin — Maltodextrin comparable in color, texture and taste to the probiotic mixture administered once a day for 3 months.
  Arms: Maltodextrin

SUMMARY:
Allergic diseases are currently one of the most important problem in medicine. Research confirms that probiotics administered during the formation of the intestinal ecosystem and the maturation of the immune system can positively influence the development of antiallergic mechanisms. The aim of the present randomized, double-blind, placebo controlled study was to evaluate the efficacy of the mixture of probiotic Lactobacillus rhamnosus ŁOCK 0900, Lactobacillus rhamnosus ŁOCK 0908, and Lactobacillus casei ŁOCK 0919 in children up to the age 2 with atopic dermatitis and food allergy to cow's milk proteins. Children received the mixture of Lactobacillus strains for 3 months every day in the daily dose of a billion bacteria or a placebo (maltodextrin). Primary outcomes included the effects of probiotic treatment on the severity of symptoms assessed with SCORing atopic dermatitis (SCORAD) index. Secondary endpoints included assessment of total IgE and selected cytokine levels. Cytokines were evaluated in supernatants obtained from peripheral blood cultures of randomly selected 20 patients from each group. The primary and secondary outcomes were assessed at 3 time points: at baseline, after the finishing the administration of probiotic/placebo, and after 9 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of atopic dermatitis according to Hanifin and Rajka criteria,
* age under 2 years (24 months)
* the SCORAD index >10
* suspected allergy to cow's milk protein

Exclusion Criteria:

* acute infections of skin,
* presence of other severe diseases
* treatment with systemic corticosteroids
* treatment with antibiotics for at least 6 weeks prior to study enrollment
* use of probiotics for the last 6 weeks prior to study enrollment

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in severity of atopic dermatitis symptoms assessed with the use the SCORAD index | From baseline at 3 months of intervention and 9 months of follow up
  The SCORAD index consists of the interpretation of the extent of the disorder (A: according to the rule of nines; 20% of the score), the intensity composed of six items (B: erythema, oedema ⁄papules, effect of scratching, oozing ⁄crust formation, lichenification and dryness; 60% of the score; each item has four grades: 0,1, 2, 3) and subjective symptoms (C: itch, sleeplessness; 20% of the score). Both subjective items are graded on a 10-cm visual analogue scale.
  The SCORAD index formula is: A ⁄5 + 7B⁄2 + C. In this formula A is defined as the extent (0-100), B is defined as the intensity (0-18) and C is defined as the subjective symptoms (0-20). The maximum SCORAD score is 103.
Changes in proportion of children with improvement or worsening of atopic dermatitis symptoms | From baseline at 3 months of intervention and 9 months of follow up
  Atopic dermatitis symptoms were assessed with the use of the SCORAD index. It was assumed that a drop >30% in the SCORAD index compared with baseline was associated with a clinically meaningful improvement. A drop<30% was associated with worsening.

SECONDARY OUTCOMES:
Changes in the level of total IgE | From baseline at 3 months of intervention and 9 months of follow up
  Total IgE level was measured using the ImmunoCap system according manufacturer's instruction.
Changes in the level of selected cytokines | From baseline at 3 months of intervention and 9 months of follow up
  The level of proinflammatory Th1 cytokines (e.g. interferon-gamma, interleukin-12), regulatory cytokines (e.g. intreleukin-10) or proallergic Th2 cytokines (e.g. interleukin-5) were measured in the supernatants obtained from the peripheral blood cultures with the use of ELISA techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Memorial Health Institute, Warsaw, Poland

REFERENCES:
- [Derived] Cukrowska B, Ceregra A, Maciorkowska E, Surowska B, Zegadlo-Mylik MA, Konopka E, Trojanowska I, Zakrzewska M, Bierla JB, Zakrzewski M, Kanarek E, Motyl I. The Effectiveness of Probiotic Lactobacillus rhamnosus and Lactobacillus casei Strains in Children with Atopic Dermatitis and Cow's Milk Protein Allergy: A Multicenter, Randomized, Double Blind, Placebo Controlled Study. Nutrients. 2021 Apr 1;13(4):1169. doi: 10.3390/nu13041169. PMID 33916192